CLINICAL TRIAL: NCT06581341
Title: Improvement of Pelvic Floor Function Using Repetitive Transcranial Magnetic Stimulation and Posterior Tibial Nerve Stimulation in Treating Neurogenic Overactive Bladder in Patients With Multiple Sclerosis
Brief Title: Enhancing Pelvic Floor Function With Transcranial Magnetic and Tibial Nerve Stimulation for Neurogenic Bladder in MS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sierra Varona SL (Other)
Collaborators: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0013; 5465 (Registry Identifier: CEIm Hospital Universitario La Princesa)
Record Dates: First submitted 2024-08-24; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Neurogenic Overactive Bladder; Multiple Sclerosis
Keywords: Múltiple Sclerosis; Neurogenic Overactive Bladder; Posterior Tibial Nerve Meuromodulation; Repetitive Transcranial Magnetic Stimulation.
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: clínical Trials with 3 arms
Who Masked: Investigator
Masking Description: This study employs a single-blind, randomized clinical trial design, with participants assigned to one of three groups: Group 1 receives repetitive transcranial magnetic stimulation (rTMS) combined with posterior tibial nerve percutaneous neuromodulation, Group 2 receives only rTMS, and Group 3 receives only posterior tibial nerve percutaneous neuromodulation. To prevent allocation bias, sealed, opaque, numbered envelopes containing color-coded cards (red for Group 1, green for Group 2, yellow for Group 3) will be used. These envelopes will be selected sequentially at the time of inclusion, ensuring that neither participants nor investigators can predict the assignments. The principal investigator will oversee randomization and administer the treatments, while the collaborating investigator, who is blinded to group assignments, will evaluate the participants. This methodology preserves the study's randomized integrity and ensures unbiased group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Combination of transcranial magnetic stimulation and percutaneous tibial nerve stimulation.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation and Percutaneous Tibial Nerve Stimulation
- Group 2 (Experimental): Repetitive Transcranial Magnetic Stimulation (rTMS):
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Group 3 (Experimental): Percutaneous tibial nerve stimulation.
  Interventions: Device: Percutaneous Tibial Nerve Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation and Percutaneous Tibial Nerve Stimulation — Repetitive Transcranial Magnetic Stimulation (rTMS): rTMS is a non-invasive procedure that uses a magnetic coil placed on the scalp to deliver magnetic pulses to the motor cortex, with the aim of improving bladder function by modulating brain activity associated with bladder control. The MagRex magnetic stimulator with an 8-shaped coil will be used at a frequency of 10 Hz, delivering 2000 pulses per session (6 seconds on, 24 seconds rest protocol) at 90% of the motor threshold. The treatment will consist of 3 sessions per week over a period of 4 weeks.
  Percutaneous Tibial Nerve Stimulation (PTNM): PTNM involves the use of electrical stimulation applied to the posterior tibial nerve to enhance bladder function by modulating neural pathways. A needle will be placed 5-6 cm proximal to the tibial malleolus, with the following parameters: 200 μs pulse duration, 20 Hz frequency, 30 minutes per session, 3 times per week for 12 weeks. The Neurotrac Pelvitone device will be used.
  Arms: Group 1
Device: Repetitive Transcranial Magnetic Stimulation — Repetitive Transcranial Magnetic Stimulation (rTMS): rTMS is a non-invasive procedure that uses a magnetic coil placed on the scalp to deliver magnetic pulses to the motor cortex, with the aim of improving bladder function by modulating brain activity associated with bladder control. The MagRex magnetic stimulator with an 8-shaped coil will be used at a frequency of 10 Hz, delivering 2000 pulses per session (6 seconds on, 24 seconds rest protocol) at 90% of the motor threshold. The treatment will consist of 3 sessions per week over a period of 4 weeks.
  Arms: Group 2
Device: Percutaneous Tibial Nerve Stimulation — Percutaneous Tibial Nerve Stimulation (PTNM): PTNM involves the use of electrical stimulation applied to the posterior tibial nerve to enhance bladder function by modulating neural pathways. A needle will be placed 5-6 cm proximal to the tibial malleolus, with the following parameters: 200 μs pulse duration, 20 Hz frequency, 30 minutes per session, 3 times per week for 12 weeks. The Neurotrac Pelvitone device will be used.
  Arms: Group 3

SUMMARY:
Multiple Sclerosis (MS) is a chronic, autoimmune, inflammatory, and degenerative neurological disorder that affects the central nervous system. Symptoms vary widely depending on the areas impacted and may include fatigue, vision issues, speech difficulties, tremors, limb weakness, loss of sensation, vertigo, coordination problems, and bladder and bowel dysfunction. Among these, lower urinary tract symptoms are particularly common and significantly impact the quality of life for MS patients.

Neurogenic overactive bladder (NOAB) is a prevalent urinary issue in individuals with MS. Treatment options for NOAB include behavioral therapy, β-3 agonists, anticholinergic agents, posterior tibial nerve neuromodulation (PTNM), botulinum toxin injections, sacral root neurostimulation, and surgical interventions.

Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation technique that may improve bladder function by modulating neural activity through an electromagnetic coil placed on the scalp. In contrast, posterior tibial nerve neuromodulation (PTNM) involves electrical stimulation of the spinal cord roots, primarily the S3 segment, to enhance bladder function.

Despite promising evidence, rTMS and PTNM are not yet widely recommended in global guidelines due to the limited number of studies, many of which are case reports. The growing prevalence of overactive bladder underscores the need for effective, non-invasive treatments to improve management and optimize current protocols.

This study aims to evaluate and compare the efficacy of rTMS and tibial nerve stimulation in managing neurogenic overactive bladder in MS patients at Hospital Universitario de la Princesa. The primary objective is to determine whether rTMS is superior, equivalent, or inferior to tibial nerve stimulation in treating NOAB.

The study's hypothesis is that the efficacy of transcranial magnetic stimulation will differ from that of tibial nerve stimulation in managing NOAB in MS patients at Hospital Universitario de la Princesa, with a focus on assessing whether rTMS offers superior, equivalent, or inferior outcomes compared to tibial nerve stimulation. This investigation seeks to provide valuable insights into the effectiveness of these treatment modalities.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic, autoimmune, inflammatory, demyelinating, and degenerative neurological disease that affects the central nervous system. Symptoms vary widely depending on the areas involved and may include fatigue, blurred vision, speech disturbances, limb weakness, tremors, loss of sensation, vertigo, coordination difficulties, and bladder and bowel dysfunctions. Among these, lower urinary tract symptoms are particularly common and significantly impact the quality of life in MS patients.

Neurogenic overactive bladder (NOAB) is the most prevalent urinary complaint in individuals with MS. Current therapeutic options for NOAB in MS include behavioral therapy, β-3 agonists, anticholinergic agents, posterior tibial nerve neuromodulation (PTNM), botulinum toxin injections, sacral root neurostimulation, and surgical interventions.

Repetitive transcranial magnetic stimulation (rTMS) is a non-invasive brain stimulation technique that may improve bladder function by modulating neural activity through an electromagnetic coil placed on the scalp. Similarly, posterior tibial nerve neuromodulation (PTNM) involves electrical stimulation of the spinal cord roots, mainly the S3 segment, to enhance bladder function.

Although current literature suggests the potential efficacy of both neuromodulation techniques for NOAB, they are not yet widely recommended in global guidelines, largely due to the limited number of studies, many of which are case reports.

The increasing incidence of overactive bladder highlights the urgent need for effective therapeutic interventions. Non-invasive neuromodulation techniques offer promising avenues to enhance treatment outcomes and optimize existing protocols.

This study aims to compare the efficacy of rTMS and tibial nerve stimulation in managing neurogenic overactive bladder in MS patients at Hospital Universitario de la Princesa. The objective is to determine whether rTMS is superior, equivalent, or inferior to tibial nerve stimulation in treating this condition.

The hypothesis posits that the efficacy of transcranial magnetic stimulation will differ from that of tibial nerve stimulation in managing NOAB in MS patients at Hospital Universitario de la Princesa, with the goal of determining whether rTMS is more effective, equally effective, or less effective than tibial nerve stimulation.

Secondary objectives include:

Assessing the efficacy of rTMS in reducing urinary symptoms associated with NOAB in MS patients.

Evaluating the combined effects of transcranial magnetic stimulation and tibial nerve stimulation on urinary symptoms.

Examining the short- and medium-term effects of the treatments on urinary symptoms.

Analyzing the impact of the treatments on the quality of life in MS patients, using the Multiple Sclerosis Quality of Life-54 Questionnaire (MsQoL-54).

Evaluating the applicability of the treatment protocols and analyzing clinical data for future neuromodulation research.

Safety and Adverse Events Monitoring

The study will adhere to current regulatory frameworks governing TMS and PTNS protocols to ensure safety and monitor adverse events. TMS is considered a well-tolerated procedure with minimal adverse effects, even in long-term studies. Commonly observed side effects, which typically resolve within a few days, include headaches, paresthesia, limb pain, restless legs syndrome, increased bladder spasticity, and nonspecific discomfort.

A review of the literature indicates no significant complications associated with percutaneous tibial nerve stimulation (PTNS). However, potential adverse events include skin irritation, increased pain at the stimulation site, rare skin lesions, allergic reactions, and general discomfort.

Any adverse events will be reported to the Ethics Committee and managed according to current safety standards, with monthly documentation. Serious adverse events will be reported immediately.

Safety Protocol

To mitigate potential risks associated with TMS and PTNS, the following safety measures will be implemented:

Proper selection of stimulation intensity and frequency. Precise location of stimulation. Application of aseptic and antiseptic techniques. Monitoring of vital signs (heart rate, blood pressure, oxygen saturation) during and after procedures to detect cardiovascular complications.

Informed consent will be obtained from participants, including comprehensive information about potential risks and the voluntary nature of participation. All personnel involved will be adequately trained in administering the techniques and identifying potential safety issues. All relevant ethical and legal regulations will be observed.

Sample Recruitment

Participants will be recruited through the Rehabilitation Physician, who will inform potential participants about the study during consultations, providing them with a Patient Information Sheet and Informed Consent Form.

Study Design

This study employs a single-blind, randomized clinical trial design. Participants will be randomly assigned to one of three groups:

Group A: rTMS combined with PTNS. Group B: rTMS alone. Group C: PTNS alone. Sealed, opaque, and numbered envelopes will be used to ensure unbiased group assignments. The anticipated start date is one month after receiving Ethics Committee approval.

Transcranial Magnetic Stimulation (TMS) Protocol

The study will use high-frequency TMS at 10 Hz, with a total of 2,000 pulses per session. The treatment duration is 30 minutes, with 12 sessions conducted over 4 weeks (3 sessions per week).

Percutaneous Tibial Nerve Stimulation (PTNS) Protocol

PTNS will involve needle placement 5-6 cm from the medial malleolus, with a pulse duration of 200 µs and a frequency of 20 Hz. Each session will last 30 minutes, with 12 sessions conducted over 4 weeks (3 sessions per week).

Randomization and Blinding

The principal investigator will conduct randomization, while the collaborating investigator will remain unaware of group assignments. The principal investigator will administer the treatments, maintaining single-blind conditions.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer Adults (Age 18-65)
* Diagnosis of Multiple Sclerosis
* Expanded Disability Status Scale (EDSS) 0-7
* Diagnosis of overactive bladder disfunction secondary to multiple sclerosis

Exclusion Criteria:

* Active urinary tract infection at the time of selection.
* Individuals with a history of urological conditions other than overactive bladder secondary to multiple sclerosis.
* Contraindications for electrical stimulation:
* Presence of metal in the skull
* Intracardiac lines
* History of increased intracranial pressure
* Significant heart disease
* Pacemaker or implantable desfibrillator usage
* Use of implanted medication pumps
* Treatment with tricyclic antidepressants or neuroleptics
* Personal or family history of epilepsy
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-01-27 (Estimated); Study Completion 2025-09-22 (Estimated)

PRIMARY OUTCOMES:
Reduction in Frequency of Urinary Urgency Episodes | Participants will complete questionnaires at four time points: 2 weeks before the start of treatment, immediately at the end of treatment, and 4 and 24 weeks post-treatment..
  Urgency urinary incontinence is marked by a sudden, intense urge to urinate, often leading to involuntary leakage. This clinical trial focuses on assessing both the presence and severity of urinary urgency in participants.It will be measured using a voiding diary. Participants will receive clear instructions on how to complete the diary, where they will record their daily voiding episodes

SECONDARY OUTCOMES:
Frequency of Urination | Participants will complete questionnaires at four time points: 2 weeks before the start of treatment, immediately at the end of treatment, and 4 and 24 weeks post-treatment.t.
  The term "frequency of urination" is defined as the number of times a person urinates within a specified time period. The frequency of urination exhibited by a participant over the course of a day is a key indicator of overall hydration status.
  The measurement of this variable is as follows: A bladder diary will be employed for the purpose of data collection. The participants will be provided with explicit instructions regarding the completion of the diary, which they will utilize to record their daily instances of urination.
Urinary Incontinence | Participants will complete questionnaires at four time points: 2 weeks before the start of treatment, immediately at the end of treatment, and 4 and 24 weeks post-treatment.
  Involuntary micturation of urine, which may manifest as dribbling, minor incontinence episodes, or significant leakage.It will be measured using a validated questionnaire, the Overactive Bladder Symptom Score (OABSS), which assesses the frequency and intensity of urinary urgency, as well as its impact on the participants' quality of life
Expanded Disability Status Scale (EDSS) | Participants will complete questionnaires at four time points: 2 weeks before the start of treatment, immediately at the end of treatment, and 4 and 24 weeks post-treatment.
  The assessment tool evaluates visual, motor, sensory, sphincteric, and cerebellar functions. The EDSS will be used to measure the effectiveness of a treatment in reducing disease progression and disability across these systems.
The Multiple Sclerosis Quality of Life-54 (MSQoL-54) Questionnaire | Participants will complete questionnaires at four time points: 2 weeks before the start of treatment, immediately at the end of treatment, and 4 and 24 weeks post-treatment.
  The 54-item questionnaire assesses multiple dimensions of quality of life, including physical function, emotional well-being, mental health, vitality, and social function. The domains deemed pertinent to this study encompass physical function, social function, and emotional well-being.
The semi-open question to assess the impact of overactive bladder on daily life. | Participants will complete questionnaires at four time points: 2 weeks before the start of treatment, immediately at the end of treatment, and 4 and 24 weeks post-treatment.
  Describe how overactive bladder symptoms affected your daily life and well-being in the past day. Include any specific instances where these symptoms significantly impacted your routine or activities.

CONTACTS AND LOCATIONS:
Overall Officials: Elena Fernández, Physiotherapist, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa

REFERENCES:
- [Background] Garcia Lopez FJ, Garcia-Merino A, Alcalde-Cabero E, de Pedro-Cuesta J. Incidence and prevalence of multiple sclerosis in Spain: a systematic review. Neurologia (Engl Ed). 2024 Oct;39(8):639-650. doi: 10.1016/j.nrleng.2022.02.004. Epub 2022 Nov 21. PMID 36410655
- [Background] Klineova S, Lublin FD. Clinical Course of Multiple Sclerosis. Cold Spring Harb Perspect Med. 2018 Sep 4;8(9):a028928. doi: 10.1101/cshperspect.a028928. PMID 29358317
- [Background] Pitt D, Lo CH, Gauthier SA, Hickman RA, Longbrake E, Airas LM, Mao-Draayer Y, Riley C, De Jager PL, Wesley S, Boster A, Topalli I, Bagnato F, Mansoor M, Stuve O, Kister I, Pelletier D, Stathopoulos P, Dutta R, Lincoln MR. Toward Precision Phenotyping of Multiple Sclerosis. Neurol Neuroimmunol Neuroinflamm. 2022 Aug 30;9(6):e200025. doi: 10.1212/NXI.0000000000200025. Print 2022 Nov. PMID 36041861
- [Background] Al Dandan HB, Coote S, McClurg D. Prevalence of Lower Urinary Tract Symptoms in People with Multiple Sclerosis: A Systematic Review and Meta-analysis. Int J MS Care. 2020 Mar-Apr;22(2):91-99. doi: 10.7224/1537-2073.2019-030. PMID 32410904
- [Background] Erden E, Ersoz M, Tiftik T, Erden E. The neurogenic bladder characteristics and treatment approaches in the patients with multiple sclerosis. Mult Scler Relat Disord. 2022 Feb;58:103439. doi: 10.1016/j.msard.2021.103439. Epub 2021 Dec 3. PMID 34954652
- [Background] Hemmett L, Holmes J, Barnes M, Russell N. What drives quality of life in multiple sclerosis? QJM. 2004 Oct;97(10):671-6. doi: 10.1093/qjmed/hch105. PMID 15367738
- [Background] Aharony SM, Lam O, Corcos J. Treatment of lower urinary tract symptoms in multiple sclerosis patients: Review of the literature and current guidelines. Can Urol Assoc J. 2017 Mar-Apr;11(3-4):E110-E115. doi: 10.5489/cuaj.4059. Epub 2017 Mar 16. PMID 28360957
- [Background] Sousa-Fraguas MC, Lastra-Barreira D, Blanco-Diaz M. Peripheral neuromodulation in women with overactive bladder syndrome: a systematic review. Actas Urol Esp (Engl Ed). 2021 Apr;45(3):177-187. doi: 10.1016/j.acuro.2020.10.003. Epub 2021 Jan 19. English, Spanish. PMID 33353738
- [Background] Canbaz Kabay S, Kabay S, Mestan E, Cetiner M, Ayas S, Sevim M, Ozden H, Karaman HO. Long term sustained therapeutic effects of percutaneous posterior tibial nerve stimulation treatment of neurogenic overactive bladder in multiple sclerosis patients: 12-months results. Neurourol Urodyn. 2017 Jan;36(1):104-110. doi: 10.1002/nau.22868. Epub 2015 Sep 9. PMID 26352904
- [Background] Martin-Garcia M, Crampton J. A single-blind, randomized controlled trial to evaluate the effectiveness of transcutaneous tibial nerve stimulation (TTNS) in Overactive Bladder symptoms in women responders to percutaneous tibial nerve stimulation (PTNS). Physiotherapy. 2019 Dec;105(4):469-475. doi: 10.1016/j.physio.2018.12.002. Epub 2018 Dec 18. PMID 30862384
- [Background] Ellaway PH, Vasquez N, Craggs M. Induction of central nervous system plasticity by repetitive transcranial magnetic stimulation to promote sensorimotor recovery in incomplete spinal cord injury. Front Integr Neurosci. 2014 May 20;8:42. doi: 10.3389/fnint.2014.00042. eCollection 2014. PMID 24904326
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Background] Centonze D, Petta F, Versace V, Rossi S, Torelli F, Prosperetti C, Rossi S, Marfia GA, Bernardi G, Koch G, Miano R, Boffa L, Finazzi-Agro E. Effects of motor cortex rTMS on lower urinary tract dysfunction in multiple sclerosis. Mult Scler. 2007 Mar;13(2):269-71. doi: 10.1177/1352458506070729. Epub 2007 Jan 29. PMID 17439897
- [Background] Pericolini M, Miget G, Hentzen C, Finazzi Agro E, Chesnel C, Lagnau P, Haddad R, Grasland M, Amarenco G. Cortical, Spinal, Sacral, and Peripheral Neuromodulations as Therapeutic Approaches for the Treatment of Lower Urinary Tract Symptoms in Multiple Sclerosis Patients: A Review. Neuromodulation. 2022 Dec;25(8):1065-1075. doi: 10.1111/ner.13525. Epub 2022 Jun 14. PMID 34496454
- [Background] Rossi S, Hallett M, Rossini PM, Pascual-Leone A; Safety of TMS Consensus Group. Safety, ethical considerations, and application guidelines for the use of transcranial magnetic stimulation in clinical practice and research. Clin Neurophysiol. 2009 Dec;120(12):2008-2039. doi: 10.1016/j.clinph.2009.08.016. Epub 2009 Oct 14. PMID 19833552
- [Background] Rossi S, Antal A, Bestmann S, Bikson M, Brewer C, Brockmoller J, Carpenter LL, Cincotta M, Chen R, Daskalakis JD, Di Lazzaro V, Fox MD, George MS, Gilbert D, Kimiskidis VK, Koch G, Ilmoniemi RJ, Lefaucheur JP, Leocani L, Lisanby SH, Miniussi C, Padberg F, Pascual-Leone A, Paulus W, Peterchev AV, Quartarone A, Rotenberg A, Rothwell J, Rossini PM, Santarnecchi E, Shafi MM, Siebner HR, Ugawa Y, Wassermann EM, Zangen A, Ziemann U, Hallett M; basis of this article began with a Consensus Statement from the IFCN Workshop on "Present, Future of TMS: Safety, Ethical Guidelines", Siena, October 17-20, 2018, updating through April 2020. Safety and recommendations for TMS use in healthy subjects and patient populations, with updates on training, ethical and regulatory issues: Expert Guidelines. Clin Neurophysiol. 2021 Jan;132(1):269-306. doi: 10.1016/j.clinph.2020.10.003. Epub 2020 Oct 24. PMID 33243615
- [Background] Finazzi-Agro E, Petta F, Sciobica F, Pasqualetti P, Musco S, Bove P. Percutaneous tibial nerve stimulation effects on detrusor overactivity incontinence are not due to a placebo effect: a randomized, double-blind, placebo controlled trial. J Urol. 2010 Nov;184(5):2001-6. doi: 10.1016/j.juro.2010.06.113. Epub 2010 Sep 20. PMID 20850833
- [Background] Tutolo M, Ammirati E, Heesakkers J, Kessler TM, Peters KM, Rashid T, Sievert KD, Spinelli M, Novara G, Van der Aa F, De Ridder D. Efficacy and Safety of Sacral and Percutaneous Tibial Neuromodulation in Non-neurogenic Lower Urinary Tract Dysfunction and Chronic Pelvic Pain: A Systematic Review of the Literature. Eur Urol. 2018 Mar;73(3):406-418. doi: 10.1016/j.eururo.2017.11.002. Epub 2018 Jan 12. PMID 29336927
- [Background] Peters KM, Carrico DJ, Perez-Marrero RA, Khan AU, Wooldridge LS, Davis GL, Macdiarmid SA. Randomized trial of percutaneous tibial nerve stimulation versus Sham efficacy in the treatment of overactive bladder syndrome: results from the SUmiT trial. J Urol. 2010 Apr;183(4):1438-43. doi: 10.1016/j.juro.2009.12.036. Epub 2010 Feb 20. PMID 20171677
- [Background] Bobes J, Bulbena A, Luque A, Dal-Re R, Ballesteros J, Ibarra N; Grupo de Validacion en Espanol de Escalas Psicometricas. [A comparative psychometric study of the Spanish versions with 6, 17, and 21 items of the Hamilton Depression Rating Scale]. Med Clin (Barc). 2003 May 17;120(18):693-700. doi: 10.1016/s0025-7753(03)73814-7. Spanish. PMID 12781095
- [Background] Keriven H, Sanchez Sierra A, Gonzalez de-la-Flor A, Garcia-Arrabe M, Bravo-Aguilar M, de la Plaza San Frutos M, Garcia-Perez-de-Sevilla G, Tornero-Aguilera JF, Clemente-Suarez VJ, Dominguez-Balmaseda D. Effects of combined treatment with transcranial and peripheral electromagnetic stimulation on performance and pain recovery from delayed onset muscle soreness induced by eccentric exercise in young athletes. A randomized clinical trial. Front Physiol. 2023 Oct 11;14:1267315. doi: 10.3389/fphys.2023.1267315. eCollection 2023. PMID 37900951
- [Background] Gutierrez-Muto AM, Bestmann S, Sanchez de la Torre R, Pons JL, Oliviero A, Tornero J. The complex landscape of TMS devices: A brief overview. PLoS One. 2023 Nov 28;18(11):e0292733. doi: 10.1371/journal.pone.0292733. eCollection 2023. PMID 38015924
- [Background] Yang DY, Zhao LN, Qiu MX. Treatment for overactive bladder: A meta-analysis of transcutaneous tibial nerve stimulation versus percutaneous tibial nerve stimulation. Medicine (Baltimore). 2021 May 21;100(20):e25941. doi: 10.1097/MD.0000000000025941. PMID 34011072
- [Background] Schwartz B, Rabinovich NR. Stimulating the development of orphan (and other) vaccines. Emerg Infect Dis. 1999 Nov-Dec;5(6):832. doi: 10.3201/eid0506.990617. No abstract available. PMID 10603222
- [Background] Kokdere F, Tirrell E, Fukuda AM, Gobin AP, Kavanaugh BC, Price LH, Carpenter LL. Do deviations from the 5 sessions per week schedule impact outcomes of transcranial magnetic stimulation for major depressive disorder? Brain Stimul. 2020 Nov-Dec;13(6):1491-1493. doi: 10.1016/j.brs.2020.08.001. Epub 2020 Aug 6. No abstract available. PMID 32768691
- See also: Guidelines. Uroweb - European Association of Urology. Retrieved September 5, 2023 — http://www.uroweb.org/guidelines/.

DOCUMENTS (1):
  • Informed Consent Form (2024-07-12): https://cdn.clinicaltrials.gov/large-docs/41/NCT06581341/ICF_000.pdf